CLINICAL TRIAL: NCT05118984
Title: Comparison Between Azithromycin vs Placebo in Cases of Meconium Stained Amniotic Fluid During the First Stage of Labor in Multigravida Women and Their Effect on Maternal and Neonatal Outcomes, a Double-blind, Placebo-controlled Randomized Clinical Trial.
Brief Title: Efficacy of Azithromycin in MSAF Cases to Improve Maternal and Neonatal Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Kamal Zaghloul, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Azithromycin in MSAF cases
Record Dates: First submitted 2021-11-05; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Meconium Stained; Azithromycin; Postpartum Endometritis
Keywords: Azithromycin; Placebo; Postpartum Endometritis
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Eligible participant will be allocated to one of two groups :
  Group 1 will be offered Azithromycin capsule (Zithromax, Pfizer) (250 mg / 12 hrs on empty stomach for 3 days).
  Group 2 will be offered placebo capsules (manufactured in pharmacy department with the same shape, colour and consistency as Azithromycin capsule for 3 days). A single pharmacist will be responsible for manufacturing of placebo capsules and packing all medications into sterile boxes and labelling of them as 1 or 2.
Who Masked: Participant, Investigator
Masking Description: Patients will be randomized to the 2 study groups according to a 2-block randomization list coded I or II at a 1:1 ratio. The randomization list will be prepared using a computer- generated random table by a statistician not otherwise involved in the study. The allocated groups will be masked in serially numbered sealed opaque envelopes that will be opened only after enrollment. Women who will be recruited give consent and open randomization envelopes in early labor, also the women will be recruited before revealing the allocation, the allocation will be blind to both the recruiter and the participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin group (Active Comparator): Azithromycin capsule (Zithromax, Pfizer) (250 mg / 12 hrs on empty stomach for 3 days).
  Interventions: Drug: Azithromycin capsule (Zithromax, Pfizer) (250 mg)
- Placebo group (Placebo Comparator): placebo capsules (manufactured in pharmacy department with the same shape, color and consistency as Azithromycin capsule every 12hrs for 3 days). A single pharmacist will be responsible for manufacturing of placebo capsules and packing all medications into sterile boxes and labelling of them as 1 or 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin capsule (Zithromax, Pfizer) (250 mg) — Azithromycin, a second generation macrolide, broad-spectrum antibacterial that stops bacterial growth by inhibiting protein synthesis and translation, treating bacterial infections Azithromycin has additional immunomodulatory effects and has been used in chronic respiratory inflammatory diseases for this purpose. .Azithromycin has been beneficial in the treatment of influenza and Middle East respiratory syndrome coronavirus (MERS-CoV) and recently has shown to be effective against severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) when used in combination with hydroxychloroquine or chloroquine.
  Arms: Azithromycin group
Drug: Placebo — A treatment that has no active properties
  Arms: Placebo group

SUMMARY:
Meconium stained amniotic fluid increases the risk of maternal complications (e.g., dystocia, operative delivery, and postpartum endometritis) and neonatal complications (e.g., sepsis, admission to the neonatal intensive care unit [NICU], and meconium aspiration syndrome). The goal of the study is to compare between Azithromycin vs Placebo in cases of meconium stained amniotic fluid during the first stage of labor in multigravida women and their effect on maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Meconium stained amniotic fluid, a troublesome situation both for obstetrician and pediatrician, it is associated with high rates of caesarean section, perinatal morbidity and mortality. The rate of meconium-stained amniotic fluid varies from 12 to 20%.It is higher in underdeveloped countries.Our study design would be a prospective randomized trial. Consented, eligible pregnant women presenting during the first stage of labor at or more than 37 weeks of gestation with meconium stained amniotic fluid will be randomized to receive Azithromycin capsule (Zithromax, Pfizer) (250 mg / 12hrs on empty stomach for 3 days)(Group 1).Group 2 will be offered placebo capsules (manufactured in pharmacy department with the same shape, color and consistency as Azithromycin capsule for 3 days).

ELIGIBILITY:
Inclusion Criteria:

1. Multigravida pregnant women with meconium stained amniotic fluid encountered either by spontaneous/artificial amniotomy during the first stage of labor in the ward provided that the gestational age at delivery is 37 weeks of gestation or more.
2. Singleton living gestation
3. Cephalic presentation
4. Adequate pelvis
5. An informed written consent for the proposed study.

Exclusion Criteria:

1. Primigravids
2. Women with previous cesarean section
3. Multifetal gestation
4. Intrauterine fetal death
5. Malpresentations
6. Prematurity (<37 weeks )
7. Abnormally invasive placenta during the current pregnancy
8. Medical disorders with pregnancy
9. Contracted pelvis
10. Evidence of maternal infection
11. Allergy to azithromycin or other macrolides that is self-reported or documented in the medical record.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Azithromycin vs Placebo in cases of meconium stained amniotic fluid during the first stage of labor in multigravida women and their effect on occurrence of maternal fever, postpartum endometritis and skin (episiotomy/tear) infection. | within 1 week from delivery
  Mothers will be followed up during her stay in the postnatal ward regarding signs of infection (fever, maternal tachycardia, offensive vaginal discharge, uterine tenderness). Postpartum follow up visit 1 week after delivery will be conducted.
Azithromycin vs Placebo in cases of meconium stained amniotic fluid during the first stage of labor in multigravida women and their effect on occurrence of neonatal fever , pneumonia and skin infection . | within 1 week from delivery
  Neonates were followed up for incidence of neonatal pneumonia, neonatal skin infection , neonatal fever.

SECONDARY OUTCOMES:
Fetal necessity for NICU admission and/or mechanical ventilation. | after delivery and within 1 week postartum
  Incidence of NICU admission and/or mechanical ventilation in neonates born to women with MSAF
Occurrence of meconium aspiration | after delivery and within 1 week postpartum
  Neonates will be followed up for presence or absence of meconium aspiration, APGAR score at 1 and 5 minutes, RDS.
2- Side effects of drug (diarrhea, stomach cramps, vomiting, allergy and anaphylactic shock). | wwithin 1 week postpartum
  Mothers follow up for incidence of side effects related to Azithromycin

CONTACTS AND LOCATIONS:
Overall Officials: Gamal GamalEldin Youssef, PHD, Study Chair — Cairo University; Eman Aly Hussein Aly, PHD, Study Director — Cairo University; Ahmed Samir Rashwan, PHD, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Cairo University, Giza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Premature Rupture of Membranes: Overview, Premature Rupture of Membranes (at Term), Premature Preterm Rupture of Membranes. Medscape. — http://emedicine.medscape.com/article/261137-overview#a2
- See also: Management of meconium-stained newborns in the delivery room. — http://doi.org/10.1891/0730-0832.37.3.141
- See also: Postpartum endometritis — http://doi.org/10.1016/j.clp.2005.04.005
- See also: What Is The Real Risk Of Infection After Waters Break? — http://www.bellybelly.com.au/birth/what-is-the-real-risk-of-infection-after-waters-break/
- See also: • American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics (2016). Practice Bulletin No. 172: Premature Rupture of Membranes. — http://doi.org/10.1097/AOG.0000000000001712
- See also: Antibiotics for meconium-stained amniotic fluid in labour for preventing maternal and neonatal infections — http://europepmc.org/backend/ptpmcrender.fcgi?accid=PMC6823264&blobtype=pdf